CLINICAL TRIAL: NCT02344615
Title: A Randomized Comparison of Nerve Stimulator and Ultrasound-guided Infraclavicular Block for Upper Extremity Surgery
Brief Title: Nerve Stimulator Versus Ultrasound-guided Infraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Chunwoo Yang, Department of Anesthesiology and pain medicine, Cheju Halla General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICB1
Record Dates: First submitted 2015-01-11; First posted 2015-01-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Pain
Keywords: nerve stimulator; ultrasound
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS-guided infraclavicular block (Active Comparator): NS-guided infraclavicular block is performed using 35 ml of 0.5% ropivacaine.
  Interventions: Procedure: NS-guided infraclavicular block
- US-guided infraclavicular block (Experimental): US-guided infraclavicular block is performed using 35 ml of 0.5% ropivacaine.
  Interventions: Procedure: US-guided infraclavicular block

INTERVENTIONS:
Procedure: NS-guided infraclavicular block — Patients received a standard single injection infraclavicular block using the lateral sagittal approach of Klaastad. The infraclavicular brachial plexus is identified using an insulated needle connected to a nerve stimulator. Placement of the needle is considered adequate if motor response of radial nerve in the hand or wrist is still present at 0.2 - 0.5mA. Ropivacaine 0.5% 35ml is used.
  Arms: NS-guided infraclavicular block
Procedure: US-guided infraclavicular block — Infraclavicular block is performed under ultrasound guidance. Linear probe is placed in a parasagittal positon below the clavicle medial to the coracoid process and adjusted to achieve a cross-sectional image of the axillary artery. Using in-plane technique, an 22-gauge insulated needle is advanced caudally and posteriorly to the axillary artery. Subsequently, 35 ml of 0.5% ropivacaine is incrementally injected.
  Arms: US-guided infraclavicular block

SUMMARY:
The investigators compared the postoperative analgesia of nerve stimulator-guided and ultrasound-guided infraclavicular block for upper extremity surgery.

DETAILED DESCRIPTION:
Ultrasound (US)-guided peripheral nerve block has increased in popularity. It has many advantages such as improved success rate, faster onset time, fewer needle passes, shorter performance time, and reduced procedural pain and vascular puncture. However, there is no information about postoperative analgesia.

Therefore, the investigators tested whether ultrasound-guided peripheral nerve block enhanced the postoperative analgesia for upper extremity surgery compared with nerve stimulator (NS) guidance.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I - III patients scheduled to undergo upper extremity surgery

Exclusion Criteria:

* coagulopathy, severe pulmonary disease, neuropathy, contralateral diaphragmatic paresis, allergy to study medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | at 24h after surgery
  time from completion of local anesthetic injection until the first request for an analgesic

SECONDARY OUTCOMES:
block performance time | at 30 min after block placement
  the time between the block needle insertion and needle withdrawal
number of needle redirections | at 30 min after block placement
  either forward or backward movement of needle at least 1 cm or more
patient discomfort | at 30 min after block placement
  pain score (0-10) during the procedure
paresthesia | at 30 min after block placement
  presence of paresthesia during the procedure
onset time | until 30min after completion of local anesthetic
  complete block of sensory nerve (radial, ulnar, median, musculocutaneous, and medial antebrachial cutaneous nerve)
motor block of hand | at 24h after surgery
  presence of motor block in the operated hand
postoperative dysesthesia | at 24h after surgery
  presence of any paresthesia in the operated extremity
supplemental analgesia | at 24h after surgery
  Rescue analgesia with 75 mg of IM diclofenac was available on demand.
Pain score | at 24h after surgery
Patient satisfaction | at 24h after surgery
  The acceptance of the anesthetic technique was evaluated using a two-point score: 1, satisfactory (if necessary, I would have the same anesthetic technique); and 2, unsatisfactory (different anesthetic technique).

CONTACTS AND LOCATIONS:
Overall Officials: Chunwoo Yang, MD, Principal Investigator — Dept. of anesthesia and pain medicine, Cheju Halla General Hospital
Locations (1):
- Cheju Halla General Hopsital, Jeju City, Jeju Self-governing Province, South Korea

REFERENCES:
- [Background] Choi S, McCartney CJ. Evidence Base for the Use of Ultrasound for Upper Extremity Blocks: 2014 Update. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):242-50. doi: 10.1097/AAP.0000000000000155. PMID 25376973
- [Background] Koscielniak-Nielsen ZJ. Ultrasound-guided peripheral nerve blocks: what are the benefits? Acta Anaesthesiol Scand. 2008 Jul;52(6):727-37. doi: 10.1111/j.1399-6576.2008.01666.x. Epub 2008 May 12. PMID 18477070